CLINICAL TRIAL: NCT05201885
Title: Oncological Differences Between Transanal and Laparoscopic Total Mesorectal Excision for Rectal Cancer.
Status: Recruiting | Type: Observational
Sponsor: Yanhong Deng (Other)
Responsible Party: Sponsor-Investigator, Yanhong Deng, Director, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Other Study IDs: GIHSYSU-22
Record Dates: First submitted 2022-01-20; First posted 2022-01-21 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-01

CONDITIONS: Rectum Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- laparoscopic surgery: Different surgical methods for rectal cancer resection
- Transanal endoscopic surgery: Different surgical methods for rectal cancer resection

SUMMARY:
The primary purpose of this study is to compare the differences of oncological in rectal cancer patients undergoing laparoscopic or transanal endoscopy radical resection. The secondary purpose is to compare the effect of two different surgical methods on prognosis.

DETAILED DESCRIPTION:
Transanal total mesorectal excision (taTME) is a new surgical procedure for total mesorectal excision (TME) by dissociating the mesorectum from the bottom through transanal endoscopic. The characteristics of TaTME are mainly summarized as transanal reverse operation, no auxiliary abdominal incision, complete mesorectal excision and specimen removal through the anus. So taTME is a natural orifice specimen extraction procedure (NOSES). However, similar to NOSES, the specific surgical approach to taTME surgery may raise oncological safety concerns. Due to the premature contact with the tumor, the squeezing of the tumor cannot be avoided during the operation. The tumor may also be squeezed when the specimen is removed through the anus, putting the tumor cells at risk of shedding into the abdominal and pelvic cavity.

Whether TaTME is safe and feasible still needs strong evidence-based medical evidence. However, there have been prospective studies related to oncological in NOSES surgery, but there is a lack of prospective clinical studies on the issue of oncological diffusion during taTME surgery. Therefore, the investigators conducted a randomized controlled study to collect the abdominal and pelvic irrigation fluids in the transanal and laparoscopic TME surgery for oncological examination, to clarify the influence of the two different surgical methods on the intraoperative oncological diffusion. The purpose of this study was to clarify the effect of two different surgical methods on intraoperative tumor cell proliferation, and to compare the long-term oncological outcomes of the two surgical methods, so as to provide more evidence-based medical evidence for the safety of taTME surgery.

ELIGIBILITY:
Inclusion Criteria:

* Primary rectal carcinoma
* Single lesion
* No metastasis

Exclusion Criteria:

* History of malignant tumors
* Acute bowel obstruction, bleeding or perforation
* Tumor over 6cm in diameter or in severe adhesion with surrounded tissues
* Severe other contradictions of surgery
* Pregnant women will be excluded

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 192 rectal cancer patients will be enrolled. Patients must be older than 18 years.
Sampling Method: Non-Probability Sample
Enrollment: 192 (Estimated)
Dates: Start 2022-01-15 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
The positive rate of oncological contamination of peritoneal washings | 1 years
  Determination of tumor cell positive rate by tumor cell examination of peritoneal washings

SECONDARY OUTCOMES:
Disease free survival | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of colorectal surgery, the Sixth Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China